CLINICAL TRIAL: NCT01284374
Title: An Investigation of Parent-son-provider Decision-making About HPV Vaccination
Brief Title: Parent-son-provider Decision-making About HPV Vaccination
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Gregory Zimet, Professor, Indiana University
Other Study IDs: Merck IISP 38094
Record Dates: First submitted 2011-01-24; First posted 2011-01-27 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Human Papillomavirus Vaccination
Keywords: HPV Vaccines; Attitude to Health; Decision Making; Qualitative Research

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Male Adolescents: Male adolescents, 13-17 years old, who are seen at community adolescent health clinics and are offered HPV vaccine
- Parents of Male Adolescents: Parents of Male Adolescents, whose adolescents are being seen at community adolescent health clinics and are offered HPV vaccine
- Health Care Providers for Males 13-17 yo: Health care providers who provide medical care to male adolescents in pediatric and adolescent clinics

SUMMARY:
The objectives of this study are:

1. To better understand factors associated with acceptance and refusal of HPV vaccine among parent-son pairs and the process of parent-son decision-making with respect to vaccination.
2. To evaluate health care providers (HCPs) attitudes, implementation intentions, and planned communication strategies with respect to HPV vaccination of adolescent boys.

Hypothesis 1: Sons will have a significant role in the process of parent-son decision-making about HPV vaccination. The relative importance of this role will increase with the son's age.

Hypothesis 2: Pediatric HCPs will be unsure about vaccinating males and will lack knowledge about issues related to male HPV infection and vaccination.

DETAILED DESCRIPTION:
This protocol will involve individual semi-structured qualitative interviews with 30 parent-son dyads and 20 pediatric health care providers. Parent-son pairs will be recruited from IUMG primary care adolescent health clinics. Recruitment will occur and consent/assent for participation obtained during the visit with the health care provider, with the physician out of the room. Interviews with parents and sons will take place after the health care appointment and after HPV vaccine acceptance/refusal. Parents and sons will be administered a brief questionnaire that will cover socio-demographic and other background information. The parent-son interviews will be separate, simultaneous one-on-one ethnographic interviews (30-60 min) that focus on the decision making process regarding HPV vaccination (yes/no). Each interview will consist of 8-10 open-ended questions, serving as an elicitation device. Sample questions include: (1) Tell me what you understand about the HPV vaccine? (2) Tell me what happened when you were in the examination room and your doctor asked you and your parent/son about getting the vaccine? (3) Was the decision made quickly, or did you have a conversation about it first? (4) Who had the most influence on the decision, you or your parent/son? (5) Why did you decide to get (or not to get) the vaccine? The interviewer will ask participants to elaborate on the meaning and contexts of their responses, and look for organization in what the participant is saying, developing and testing hypotheses during the interview. Each interview will be conducted by a trained, gender-matched research assistant.

Health care providers will be interviewed at a different time, and the interviews (25-30 min) will focus on HPV vaccine related attitudes, supply, costs, communication and perceived benefits associated with vaccinating adolescent males, rather than care to specific patients. Sample questions include: (1) How do you inform patients about the HPV vaccine? (2) What is the specific wording that you use when you offer HPV vaccine? Be very specific. Don't leave out any detail.

ELIGIBILITY:
Inclusion Criteria:

Adolescent:

* English-speaking adolescent boys
* 13-17 years of age
* No prior receipt of HPV vaccine
* Accompanied by parent

Parent:

* English-speaking or Spanish-speaking parent

Health Care Provider:

* Physician
* Provides care to adolescent boys 13-17 years of age

Exclusion Criteria:

Adolescent:

* Non-English-speaking
* Younger than 13 or older than 17
* Previous receipt of 1 or more doses of HPV vaccine

Parent:

* Non-English-speaking and Non-Spanish-speaking

Health Care Provider:

* Not a physician
* Does not provide care to males 13-17 years of age

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parent-Adolescent pairs attending community-based adolescent health primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Decision Regarding Acceptance/Refusal of 1st Dose of HPV Vaccine | Up to 1 hour
  The semi-structured interviews with parents & sons will focus on how the decision was made to accept or refuse HPV vaccine. The interviews will take place immediately after the clinic visit during which the vaccination decision was made.
Health care providers decision-making regarding HPV vaccination of males | Up to 1 hour
  Semi-structured interviews will be conducted with 20 health care providers regarding their decision-making around vaccinating adolescent male patients against HPV

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Zimet, PhD, Principal Investigator — Indiana University
Locations (1):
- IU Medical Group Primary Care Clinic (IUMG-PC), including Wishard primary care clinics, Indianapolis, Indiana, United States